CLINICAL TRIAL: NCT02226315
Title: A Retrospective Analysis of Fetal Outcome Compared to Massively Parallel Sequencing Test Results Obtained From Multiple Gestation Pregnancies at Increased Risk for Fetal Chromosomal Aneuploidy
Brief Title: Clinical Performance of the MaterniT21 PLUS LDT in Multiple Gestation Pregnancies
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment of eligible subjects
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: SQNM-T21-109
Record Dates: First submitted 2014-08-20; First posted 2014-08-27 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Down Syndrome; Edwards Syndrome; Patau Syndrome; Turner Syndrome
Keywords: noninvasive prenatal testing
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Turner Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Some subjects will be asked to provide a buccal cell sample for sequencing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple gestations: Women with a multiple gestation who were evaluated with the MaterniT21 PLUS LDT and have passed their Estimated Date of Delivery (EDD).

SUMMARY:
This study will evaluate the clinical performance of massively parallel sequencing (MPS) using the MaterniT21 PLUS LDT in the detection of fetal aneuploidy in circulating cfDNA extracted from a maternal blood sample obtained from women pregnant with a multiple gestation who were at increased risk for fetal aneuploidy.

ELIGIBILITY:
Inclusion Criteria:

* Subject was pregnant with a multiple gestation and received NIPT with the MaterniT21 PLUS LDT and a valid test result is available;
* Subject was 18 years of age or older at the time of NIPT;
* Subject provides signed and dated informed consent in English;

Exclusion Criteria:

* Subjects' treating physician is not located in the United States.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a multiple gestation who were evaluated with the MaterniT21 PLUS LDT and have passed their Estimated Date of Delivery (EDD).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Clinical Performance (Sensitivity/Specificity) of MaterniT21 PLUS LDT Assay | Subjects contacted within 3 years after pregnancy is completed
  Results of the MaterniT21 PLUS LDT will be compared to the pregnancy outcome data obtained from the patient

CONTACTS AND LOCATIONS:
Overall Officials: Richard Porreco, MD, Principal Investigator — Presbyterian/St. Luke's Medical Center
Locations (1):
- Presbyterian/St. Luke's Medical Center, Denver, Colorado, United States